CLINICAL TRIAL: NCT03707080
Title: DAA-PASS: A Post-Authorisation Safety Study of Early Recurrence of Hepatocellular Carcinoma in HCV-Infected Patients After Direct-Acting Antiviral Therapy
Brief Title: Direct Acting Antiviral-Post Authorization Safety Study
Status: Completed | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-HCC DAA-PASS
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-05

CONDITIONS: Hepatitis C; Hepatocellular Carcinoma
MeSH Terms: conditions — Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: The prospective DAA-PASS cohort will include a subset of HCV RNA positive participants in the TARGET-HCC study who meet entry criteria including hepatitis C (with no prior history of DAA therapy) and newly diagnosed Barcelona Clinic Liver Cancer (BCLC) Stage A HCC.
  Participants will be enrolled in the countries participating in TARGET-HCC which will include: United States (US), France, Germany, Italy, and Spain.
- Historical: The historical cohort will be derived from the ITA.LI.CA database, which includes data on all consecutive patients with HCC who were managed within participating centers in Italy. The historical cohort will include patients from the ITA.LI.CA database who have active HCV infection who were not treated for HCV (IFN-based or DAA-based regimens) during the followup period, with initial HCC diagnosis BCLC Stage A, and subsequent successful treatment of HCC with curative therapy.

SUMMARY:
This is an independent optional sub-study parallel to TARGET-HCC (NCT02954094). The purpose of Direct-Acting Antiviral-Post Authorization Safety Study (DAA-PASS) is to investigate the impact of exposure to direct-acting antivirals (DAAs) on early recurrence of hepatocellular carcinoma (HCC) in hepatitis C virus (HCV)-infected patients following successful HCC treatment interventions.

ELIGIBILITY:
Screening Inclusion Criteria:

* Current participant in TARGET-HCC
* Adults, age ≥18 years
* First diagnosis of HCC (mixed HCC/cholangiocarcinoma may be included). Diagnosis may be histological/cytological and/or radiological.
* BCLC Stage A
* Underwent, undergoing, or planned to undergo therapy for HCC, with exception that transplant as prior or planned treatment for HCC is excluded.
* HCV RNA positive

Screening Exclusion Criteria:

* Inability to provide informed consent
* HCC-free imaging (as defined in Section 9.1.1) after treatment of initial HCC prior to Screening (see Section 9.2.9 for imaging details)
* Prior liver transplantation
* Hepatitis B Virus (HBV) surface antigen positive (HBsAg)
* Previously treated with direct-acting antiviral agents (not DAA-naïve); Note that prior (peg)IFN and/or ribavirin therapy is allowed

Enrollment Inclusion Criteria:

* Continued participation in TARGET-HCC
* No recurrence or progression of initial HCC beyond BCLC Stage A prior to Enrollment/Baseline
* HCC-free imaging (as defined in Section 9.1.1) at Enrollment/Baseline (see Section 9.2.9 for imaging details; participants may remain in Screening until an HCC-free image is obtained)
* Remains DAA-naïve (prior therapy with (peg)IFN and/or ribavirin is allowed)

Enrollment Exclusion Criteria:

- Liver transplantation since Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective DAA-PASS cohort will include a subset of HCV RNA positive participants in the TARGET-HCC study who meet entry criteria including hepatitis C (with no prior history of DAA therapy) and newly diagnosed Barcelona Clinic Liver Cancer (BCLC) Stage A HCC. Participants will be enrolled in the countries participating in TARGET-HCC which will include: United States (US), France, Germany, Italy, and Spain.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Time to HCC recurrence - Prospective Cohort | up to 24 months
  Time to HCC recurrence associated with DAA therapy relative to no DAA therapy in the prospective cohort.

SECONDARY OUTCOMES:
Number of events of early HCC recurrence - Prospective Cohort | up to 24 months
  Number of events (early HCC recurrence) associated with DAA therapy relative to no DAA therapy in the prospective cohort.
Time to HCC recurrence - Prospective Cohort relative to Historical Cohort | up to 24 months
  Time to HCC recurrence associated with DAA therapy in the prospective cohort relative to no DAA therapy in the historical cohort.
Number of events of early HCC recurrence - Prospective Cohort relative to Historical Cohort | up to 24 months
  Number of events (early HCC recurrence) associated with DAA therapy in the prospective cohort relative to no DAA therapy in the historical cohort.
  historical cohort of HCV patients not exposed to DAA with initial HCC diagnosis and subsequent successful treatment of HCC.

CONTACTS AND LOCATIONS:
Locations (61):
- United States (46):
  - Banner University Medical Center, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California - Davis Clinical Trials, Sacramento, California
  - University of California - San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Gastro Florida, Clearwater, Florida
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - University of Florida - Health Gastroenerology, Jacksonville, Florida
  - Schiff Center for Liver Diseases, Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Division of Gastroenterology and Hepatology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Northwell Health - Center for Liver Disease, Manhasset, New York
  - New York University Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolinas HealthCare System Center for Liver Disease, Charlotte, North Carolina
  - Providence Health & Services Cancer Clinical Trials, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center - GI Research Office, Nashville, Tennessee
  - Clinical Research Institute@ Methodist Dallas Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott & White All Saints, Fort Worth, Texas
  - Research Specialists of Texas, Houston, Texas
  - University of Virginia Transplant Center, Charlottesville, Virginia
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- France (2):
  - CHU de Nice - Hôpital L'Archet 2, Nice
  - Hôpitaux Universitaires Paris Centre, Paris
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
- Italy (4):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - A.O.U.P. di Palermo, Palermo
  - Humanitas Mirasole IRCCS, Rozzano
  - IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo
- Spain (5):
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No